CLINICAL TRIAL: NCT03999489
Title: Study of the Psychometric Properties and a Measure of Utility Determinants ( the SF- 6D) in Patients With Early Inflammatory Low Back Pain
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/CGV-01
Record Dates: First submitted 2016-09-12; First posted 2019-06-26 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Spondylarthritis
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The general main objective of our study is to investigate the psychometric properties, the levels and determinants of the extent of SF- 6D utility in patients followed for recent back pain inflammatory disease.

The specific objectives are :

* Study the feasibility of the tool considering missing data, distribution, construct validity, reproducibility, sensitivity to change or clinically different groups (discriminative ability) the extent of SF -6D utility .
* Study the impact of socio-demographic characteristics, disease characteristics and quality of life, comorbidities at baseline on the measurement of utility and sensitivity to change.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be given free and informed consent and signed the consent

  * The patient must be affiliated or beneficiary of a health insurance plan
  * patients aged 18 years and under 50
  * inflammatory back pain (buttocks , lumbar or thoracic spine )
  * fulfilling the criteria of Calin or Berlin (30,31)
  * duration of symptoms than three months and less than three years
  * symptoms suggestive of spondyloarthritis as assessed by the local investigator ( score≥5 on a numerical scale from 0 to 10 where 0 = no evocative and 10 = very suggestive of spondyloarthritis ) .

Exclusion Criteria:

* Another clearly defined spinal disease (eg discarthrose )

  * history of treatment with biotherapy
  * taking glucocorticoids allowed only in low dose of less than 10mg of prednisone daily and stable for at least four weeks before inclusion
  * Current or history anomalies that could interfere with the validity of informed consent and / or prevent a patient's optimal adhesion to the cohort (eg , alcoholism , mental illness) .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 708 patients with early inflammatory low back pain included in the French cohort DESIR
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Level of utility measured by the SF-6D | baseline (0 months)
  The SF-6D derives from 11 questions of the SF36 using the algorithm of Brazier et al which then provides a unique score. It has 6 dimensions: Physical Function, Role Limitation, Social Function, Pain, Mental Health and Vitality with 4 to 6 levels of responses depending on the dimension. SF-6D thus makes it possible to describe 18,000 health conditions. The utility score obtained with SF-6D varies between 0.29 and 1.
Level of utility measured by the SF-6D | 6 months
  The SF-6D derives from 11 questions of the SF36 using the algorithm of Brazier et al which then provides a unique score. It has 6 dimensions: Physical Function, Role Limitation, Social Function, Pain, Mental Health and Vitality with 4 to 6 levels of responses depending on the dimension. SF-6D thus makes it possible to describe 18,000 health conditions. The utility score obtained with SF-6D varies between 0.29 and 1.
Level of utility measured by the SF-6D | 12 months
  The SF-6D derives from 11 questions of the SF36 using the algorithm of Brazier et al which then provides a unique score. It has 6 dimensions: Physical Function, Role Limitation, Social Function, Pain, Mental Health and Vitality with 4 to 6 levels of responses depending on the dimension. SF-6D thus makes it possible to describe 18,000 health conditions. The utility score obtained with SF-6D varies between 0.29 and 1.

IPD SHARING:
Plan to Share IPD: No